CLINICAL TRIAL: NCT00856908
Title: A Randomised, Single-Blind, Placebo-Controlled, Phase IIa Study to Assess the Safety and Tolerability After Multiple Oral Doses of AZD1656 During Four Weeks in T2DM Subjects Treated With Insulin
Brief Title: Safety and Tolerability After Four Weeks of Treatment With AZD1656 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1020C00020
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2012-11-26 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-11

CONDITIONS: Type II Diabetes
Keywords: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD1656

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Dose titration of oral suspension during 4 days to a tolerable dose given twice daily. Subjects will thereafter be treated with this dose twice daily for another 24 days
  Interventions: Drug: AZD1656
- 2 (Placebo Comparator): Dose titration of oral suspension during 4 days to a tolerable dose given twice daily. Subjects will thereafter be treated with this dose twice daily for another 24 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1656 — Tolerable dose given twice daily
  Arms: 1
Drug: Placebo — Tolerable dose given twice daily
  Arms: 2

SUMMARY:
The purpose of this study is to assess the 1 month safety and tolerability after multiple oral doses of AZD1656 in patients with Type 2 Diabetes Mellitus Treated with Insulin

ELIGIBILITY:
Inclusion Criteria:

* type II diabetes patients, female with non child-bearing potential
* Subjects with T2DM diagnosis for at least one year, treated with insulin alone or insulin in combination with other anti-diabetic drugs. Subjects must have been treated with insulin the last 3 months prior to enrolment (screening)
* HbA1c <11% at enrolment (screening) (HbA1c value according to international Diabetes Control and Complications Trial [DCCT] standard).
* FPG in the range of 7.0 to 13.0 mmol/L (126 to 234 mg/dL)

Exclusion Criteria:

* History of ischemic heart disease, symptomatic heart failure, stroke, transitory ischemic attack or symptomatic peripheral vascular disease
* Use of glitazones, warfarin, amiodarone within 3 months prior to enrolment (screening) and use of potent CYP450 inhibitors, eg, ketoconazole and macrolide antibiotics within 14 days before randomisation.
* Any clinically significant abnormality identified on physical examination, laboratory tests or ECG, which in the judgment of the investigator would compromise the patients' safety or successful participation in the clinical study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, PhD, Prof., Study Director — AstraZeneca R&D Mölndal; Marcus Hompesch, MD, Principal Investigator — Profil Institut for Clinical Research Inc.
Locations (1):
- Research Site, Chula Vista, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: AZD1656 dose titration of oral suspension during 4 days to a tolerable dose given twice daily. Subjects will thereafter be treated with this dose twice daily for another 24 days
- Placebo Comparator: placebo Dose titration of oral suspension during 4 days to a tolerable dose given twice daily. Subjects will thereafter be treated with this dose twice daily for another 24 days
Period: Overall Study
Arm/Group | Experimental | Placebo Comparator
Started | 15 | 5
Completed | 14 | 5
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Placebo Comparator | Total
Number analyzed (Participants) | 15 | 5 | 20
Age Continuous [Mean (Full Range); unit: years] | 52.6 [40 to 65] | 57.2 [41 to 69] | 53.8 [40 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure, Change From Baseline to End of Treatment
Time Frame: Baseline is pre-dose first day of dosing, end of treatment is the morning following the treatment period
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 14 | 5
mmHg | 0.4 (8.5) | 5.0 (6.4)

2. Primary Outcome: Diastolic Blood Pressure, Change From Baseline to End of Treatment
Time Frame: Baseline is pre-dose first day of dosing, end of treatment is the morning following the treatment period
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 14 | 5
mmHg | 3.4 (7.6) | 0.6 (2.9)

3. Primary Outcome: Pulse, Change From Baseline to End of Treatment
Time Frame: Baseline is pre-dose first day of dosing, end of treatment is the morning following the treatment period
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 14 | 5
beats/min | 0.7 (4.4) | -5.4 (4.0)

4. Primary Outcome: Weight, Change From Baseline to End of Treatment
Time Frame: Baseline is the day before first dose, end of treatment is last day of treatment
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 14 | 5
kg | -0.54 (1.65) | -1.32 (1.18)

5. Primary Outcome: Clinically Relevant Change of Laboratory Variables
Description: Number of participants with clinically relevant change of laboratory variables (clinical chemistry, haematology and urinalysis parameters
Time Frame: Measured regularly from day before first dose to day after last dose
Measure: Number; unit: Participants
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 15 | 5
Participants | 0 | 0

6. Secondary Outcome: Area Under the Plasma Concentration vs Time Curve (AUC0-24) of AZD1656
Description: Dose-adjusted to a total daily dose of 100 mg due to titrated doses
Time Frame: Measured last day of treatment
Measure: Geometric Mean (95% Confidence Interval); unit: umol*h/L
Arm/Group | Experimental
Number analyzed (Participants) | 14
umol*h/L | 23.49 [18.73 to 29.45]

7. Secondary Outcome: Maximum Plasma Concentration of AZD1656
Description: Dose-adjusted to a morning dose of 50 mg due to titrated doses
Time Frame: Measured following the morning dose last day of treatment
Measure: Geometric Mean (95% Confidence Interval); unit: umol/L
Arm/Group | Experimental
Number analyzed (Participants) | 14
umol/L | 2.415 [1.992 to 2.928]

8. Secondary Outcome: Time to Reach Maximum Plasma Concentration of AZD1656
Time Frame: Measured last day of treatment
Measure: Median (Full Range); unit: h
Arm/Group | Experimental
Number analyzed (Participants) | 14
h | 0.500 [0.25 to 2.50]

9. Secondary Outcome: Terminal Elimination Half-life of AZD1656
Time Frame: Measured following the evening dose last day of treatment
Measure: Mean (Full Range); unit: h
Arm/Group | Experimental
Number analyzed (Participants) | 13
h | 5.239 [3.10 to 10.1]

10. Secondary Outcome: Apparent Oral Clearance of AZD1656
Time Frame: Measured last day of treatment
Measure: Mean (Full Range); unit: L/h
Arm/Group | Experimental
Number analyzed (Participants) | 14
L/h | 9.382 [4.92 to 16.2]

11. Secondary Outcome: P-Glucose (AUC0-24)/24, Change From Baseline to End of Treatment
Description: Log ratio (End of treatment/Baseline) has been analysed in an ANCOVA model, using treatment as fixed factor and log(Baseline) as covariate. Resulting estimates have been back-transformed from the log-scale and then multiplied by 100 to obtain the relative ratio (end of treatment/placebo) in percent. Changes in percent have been obtained by subtraction by 100.
Time Frame: Baseline is the day before first dose, end of treatment is last day of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: relative change in percent
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 14 | 5
relative change in percent | -7 [-19 to 6.2] | 4 [-18 to 33]

12. Secondary Outcome: S-Insulin (AUC0-24)/24, Change From Baseline to End of Treatment
Description: as for outcome 11
Time Frame: Baseline is the day before first dose, end of treatment is last day of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: relative change in percent
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 14 | 5
relative change in percent | -2 [-15 to 12] | -29 [-45 to -9.3]

13. Secondary Outcome: S-C-Peptide (AUC0-24)/24, Change From Baseline to End of Treatment
Description: as for outcome 11
Time Frame: Baseline is the day before first dose, end of treatment is last day of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: relative change in percent
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 14 | 5
relative change in percent | -4 [-18 to 13] | -3 [-26 to 28]

ADVERSE EVENTS:
Arm/Group | Experimental | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/5
Other Adverse Events (participants affected / at risk) | 13/15 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=15) | Placebo Comparator (N=5)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 1
Application Site Reaction (Injury, poisoning and procedural complications) | 2 | 0
Catheter Site Pain (Injury, poisoning and procedural complications) | 2 | 0
Blood Glucose Decreased (Investigations) | 2 | 0
Iron Deficiency Anaemia (Metabolism and nutrition disorders) | 0 | 1
Oedema Peripheral (Metabolism and nutrition disorders) | 1 | 0
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 | 0
Headache (Nervous system disorders) | 10 | 1
Restless Legs Syndrome (Nervous system disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ecchymosis (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The primary objective of the study was to assess safety and tolerability and hence the study was not sized based on statistical considerations. The most import outcome, "no safety or tolerability concerns were identified", is not a numerical variable

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CONTRACT RESEARCH ORGANIZATION AGREEMENT by and between ASTRAZENECA AB and the CRO. CRO agrees that AstraZeneca shall have the exclusive right to publish the results of the Study, including all Work Product, and that such results may not be published or otherwise disseminated by CRO without the prior written approval of AstraZeneca.